CLINICAL TRIAL: NCT01643265
Title: Effect of Whey and Albumin Protein on Plasma Levels of Amino Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MTI2012-CS02
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Healthy Men and Women

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whey Milk Protein (Active Comparator)
  Interventions: Dietary Supplement: Whey Milk Protein
- Bovine Albumin Concentrate (Experimental)
  Interventions: Dietary Supplement: Bovine Albumin Concentrate

INTERVENTIONS:
Dietary Supplement: Whey Milk Protein — 20 grams of Whey Milk Protein
  Arms: Whey Milk Protein
Dietary Supplement: Bovine Albumin Concentrate — 20 grams of Bovine Albumin Concentrate
  Arms: Bovine Albumin Concentrate

SUMMARY:
The purpose of this study will allow us to examine how quickly and to what extent plasma amino acids levels rise after ingesting a single dose of either whey or albumin protein. The investigators anticipate that the amino acids from albumin concentrate protein will rise as quickly and to the same extent as amino acids from whey protein. These findings will help us to understand the biological availability of these proteins and efficacy of the supplement so that consumers may be presented with nutritional options.

ELIGIBILITY:
Inclusion Criteria:

* normal Healthy volunteers
* free of serious illness/disease such as hypertension, kidney or liver disease

Exclusion Criteria:

* taking dietary protein or amino acid supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Amino acid concentration | 210 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rick Sharp, PhD, Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Ames, Iowa, United States